CLINICAL TRIAL: NCT01283061
Title: An Open Label, Balanced, Randomized, Two-Treatment, Two-Period, Two-Sequence, Single Dose, Crossover, Bioavailability Study Of Zafirlukast Tablets 20 mg of Dr. Reddy's Laboratories Limited, India Comparing With That of 'ACCOLATE' Tablets 20 mg of Astrazeneca Pharmaceuticals, USA In Healthy Adult Human Subjects Under Fasting Conditions.
Brief Title: Bioequivalence Study of Zafirlukast Tablets 20 mg of Dr. Reddy's Laboratories Limited Under Fasting Condition
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Dr. Reddy's Laboratories Limited (Industry)
Responsible Party: Director-Research & Development, Dr. Reddy's Laboratories Limited
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: BA0759156
Record Dates: First submitted 2011-01-24; First posted 2011-01-25 (Estimated); Last update posted 2011-01-26 (Estimated); Status verified 2011-01

CONDITIONS: Healthy
MeSH Terms: interventions — zafirlukast

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- zafirlukast (Experimental): Zafirlukast Tablets 20 mg of Dr. Reddys Laboratories Limited
  Interventions: Drug: Zafirlukast
- Accolate (Active Comparator): ACCOLATE tablets manufactured by IPR pharmaceuticals and manufactured for Astrazeneca Pharmaceuticals
  Interventions: Drug: Zafirlukast

INTERVENTIONS:
Drug: Zafirlukast — Zafirlukast tablets 20 mg
  Other Names: Accolate tablets 20 mg

SUMMARY:
The objective of this study was to compare the relative bioavailability of zafirlukast tablets 20 mg with that of 'ACCOLATE®' tablets 20 mg (zafirlukast tablets 20 mg) in healthy, adult, human, subjects under fasting conditions and to monitor safety of subjects.

DETAILED DESCRIPTION:
open label, randomized, two-period, two treatment, two sequence, crossover, balanced single dose comparative oral bioavailability study in healthy, adult, human subjects under fasting conditions.44 healthy, adult, human subjects.There was 11-day interval between treatments.

ELIGIBILITY:
Inclusion Criteria:

1. The subjects should be healthy human between 18 and 45 years.
2. The subjects should be screened within 21 days prior to the administration of first dose of the study drug.
3. The subjects should have a BMI between 18.5 and 24.9 weight in kg/ height2 in meter.
4. The subjects should be able to communicate effectively with study personnel.
5. The subjects should be able to give written informed consent to participate in the study.

   If subject is a female volunteer and
6. Is of child bearing potential practicing an acceptable method of birth control for the duration of the study as judged by the investigator(s), such as condoms,foams, jellies, diaphragm, intrauterine device (IUD), or abstinence.
7. Is postmenopausal for at least 1 year.
8. Is surgically sterile (bilateral tubal ligation, bilateral oophorectomy, or hysterectomy has been performed on the subject).

Exclusion Criteria:

1. The subjects who have a history of allergic responses to zafirlukast or other related drugs.
2. The subjects who have used enzyme-modifying drugs within 30 days prior to receiving the first dose of study medication.
3. The subjects who have history of drug dependence, recent history of alcoholism or of moderate alcohol uses.
4. The subjects who have significant diseases or clinically significant abnormal findings during screening, medical history, physical examination, laboratory evaluations, ECG and X-ray recordings.
5. The subjects who have any disease or condition which might compromise the haemopoietic, gastrointestinal, renal, hepatic, cardiovascular, respiratory, central nervous system, diabetes, psychosis or any other body system.
6. The subjects who have a history or presence of bronchial asthma
7. The subjects who are smokers who smoke more than or equal to 10 cigarettes per day or more than or equal to 20 biddies per day or those who cannot refrain from smoking during study period.
8. The subjects with a history of difficulty with donating blood or difficulty in accessibility of veins.
9. The subjects who have donated 1 unit (350 ml / 450 ml) blood within 90 days prior to receiving the first dose of study medication.
10. The subjects who have a positive hepatitis screen (includes subtypes A, B, C and E)
11. The subjects who have a positive test result for HIV antibody and / or syphilis(RPR/VDRL).
12. The subject who receives an investigational product, or has participated in a drug research study within a period of 90 days prior to the first dose of the study medication administration.
13. Female volunteers demonstrating a positive pregnancy screen.
14. Female volunteers who are currently breast-feeding.
15. Female volunteers not willing to use contraception during the study.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 44 (Actual)
Dates: Start 2007-12; Primary Completion 2008-01 (Actual); Study Completion 2008-01 (Actual)

PRIMARY OUTCOMES:
Bioequivalence on Cmax and AUC parameters | 13 days

CONTACTS AND LOCATIONS:
Overall Officials: Ronak Modi, MBBS, Principal Investigator — BA Research India Ltd.
Locations (1):
- BA Research India Ltd., Ahmedabad, Bodakdev, India